CLINICAL TRIAL: NCT05314361
Title: Online Public Health Nurse Delivered 1-Day Cognitive Behavioural Therapy (CBT)-Based Workshops for Postpartum Depression Symptoms: Pilot Study
Brief Title: Public Health Nurse-Delivered 1-Day CBT Workshops Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHN1DayCBTPilot
Record Dates: First submitted 2022-03-21; First posted 2022-04-06 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: A parallel-group Ontario-wide RCT with experimental (workshop) and TAU (control) groups will address our objectives. Participants will be randomly assigned in a 1:1 ratio to the treatment or control groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and the research coordinator cannot be blinded to group condition though the research assistants making reminder calls and data analysts will not be aware of group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment - 1 Day CBT-Based Workshop (Experimental): Participants assigned to the treatment arm will attend a day long CBT-based workshop delivered by two trained public health nurses in addition to receiving usual care.
  Interventions: Behavioral: 1-Day Cognitive Behavioural Therapy-Based Workshop
- Control - usual care (No Intervention): Participants assigned to the control arm will continue to receive standard postnatal care from their healthcare providers.

INTERVENTIONS:
Behavioral: 1-Day Cognitive Behavioural Therapy-Based Workshop — The Online Workshop is a day-long intervention delivered by two trained public health nurses consisting of 6 hours of instruction delivered in 4 modules. The 1st contains information on PPD etiology with a focus on modifiable cognitive risk factors (e.g., negative thoughts, maladaptive core beliefs). The 2nd module focuses on cognitive skills including cognitive restructuring. The 3rd builds behavioural skills such as problem solving, behavioural activation, assertiveness, sleep strategies, and using supports. The final module provides an opportunity for goal setting/action planning. Teaching methods include didactic sections, group exercises, and role-plays. Regular breaks are incorporated. Each participant is given a professionally designed manual to facilitate learning. We also provide a list of region-specific PPD resources and a copy of the Canadian Practice Guidelines for the treatment of PPD (written by the NPA).
  Arms: Treatment - 1 Day CBT-Based Workshop

SUMMARY:
Public Health Nurses received training to deliver a day-long Cognitive Behavioural Therapy-based workshop for treating postpartum depression. Participants in the study are randomly assigned to the treatment group (1-day CBT workshop) or control group (usual postnatal care). Data will be collected from all participants at baseline, 3 and 6 months.

The study will aim to assess the feasibility of our methods and estimate the treatment effect of the primary outcome in preparation for a larger RCT. Objectives include:

* Recruit and randomize 96 participants within 5 months
* Questionnaire completion - 75% of participants complete all three questionnaires and structured interviews
* Retention - 75% of participants remain in study until completion
* 75% of participants in treatment group complete the intervention
* Estimate treatment effect and variance

DETAILED DESCRIPTION:
Postpartum depression (PPD) is one of the most common complications of childbirth, affecting 1 in 5 mothers. Left untreated, it increases the risk of future depressive episodes and can have profound effects on offspring. A single case of PPD has been estimated to cost as much as $150,000 over the lifespan, or $3 billion for each annual cohort of Canadian births.

Current clinical practice guidelines (including those written by the NPA) recommend evidence-based psychotherapies (e.g., cognitive behavioural therapy (CBT)) as 1st-line treatments for the vast majority of mothers with PPD. The key role that psychotherapy plays in the treatment of PPD is further emphasized by the US Preventive Services Task Force which recommends universal PPD screening, but "only when CBT or other evidence-based counseling is available."

While treating PPD can reduce its adverse effects, safe, timely, accessible interventions are essential to optimizing outcomes. However, only treatments that can be upscaled can have an impact on PPD at the population level.

The delivery of psychotherapy in large groups (up to 30 participants) is a relatively new phenomenon, but may be capable of addressing mothers' needs, as well as treating PPD on the scale required to address its prevalence. Brief (i.e., 1-Day) interventions contain the core content of more comprehensive, evidence-based interventions, but their brevity makes them easier to disseminate beyond traditional treatment settings (e.g., in public health). 1-Day CBT-Based Workshops have been delivered by trained mental health professionals (psychologists, psychiatrists) to treat generalized anxiety disorder and depression in general population samples, and postpartum depression.

The purpose of this pilot study is to determine the feasibility of our study procedures and estimate the treatment effect and variance of the primary outcome in preparation for a larger RCT to determine the effectiveness of a Public Health Nurse-Delivered 1-Day Cognitive Behavioural Therapy-Based Workshop for postpartum depression.

A parallel-group Ontario-wide RCT with experimental (workshop) and TAU (control) groups will address our objectives. Participants in both groups will complete all study questionnaires and be compared at baseline, and 3 and 6 months.

The experimental group will receive the Online 1-Day workshop (delivered by 2 PHNs) in addition to TAU, and the control group will receive TAU alone.

Participants will be mothers who have an infant under 12 months, who are 18 years or older, who are experiencing elevated symptoms of postpartum depression and who are free of current bipolar, psychotic and/or substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have infant <12 months at time of recruitment
* fluent in written/spoken English

Exclusion Criteria:

* current bipolar, psychotic and/or substance use disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited in recruitment period | 5 months
  Recruit and randomize 96 participants within 5 months (48 treatment into four 1-day workshops (12 per workshop) and 48 control)
Number of participants who complete all data collection procedures | 6 months
  75% of participants complete all data collection procedures at all time points
Number of participants who complete study (retention) | 6 months
  75% of participants remain enrolled in the study until completion
Number of participants who complete the intervention (adherence) | 6 months
  75% of participants who are enrolled in the treatment group will complete the 1-Day CBT-based workshop

SECONDARY OUTCOMES:
Estimate Treatment effect - Edinburgh Postnatal Depression Scale (EPDS) | 3 months
  Estimate treatment effect of primary outcome for later RCT - The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score ≥13 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change.

OTHER OUTCOMES:
GAD-7 | 3 months
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) (32) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. Items are scored on a 4-point scale from 0 to 3, with a higher score indicating an increased risk of GAD. A cutoff of ≥11 defines clinically important levels of anxiety symptoms.
GAD-7 | 6 months
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) (32) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. Items are scored on a 4-point scale from 0 to 3, with a higher score indicating an increased risk of GAD. A cutoff of ≥11 defines clinically important levels of anxiety symptoms.
Multidimensional Scale of Perceived Social Support (MSPSS) | 3 months
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Multidimensional Scale of Perceived Social Support (MSPSS) | 6 months
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Parenting Stress Index (PSI-SF) | 3 months
  The Parenting Stress Index (short form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
Parenting Stress Index (PSI-SF) | 6 months
  The Parenting Stress Index (short form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
The Postpartum Bonding Questionnaire (PBQ) | 3 months
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
The Postpartum Bonding Questionnaire (PBQ) | 6 months
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 3 months
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 6 months
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
EQ-5D-5L | 3 months
  A utility-based health-related quality of life self-report instrument consisting of five questions covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach).
EQ-5D-5L | 6 months
  A utility-based health-related quality of life self-report instrument consisting of five questions covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach).
Healthcare Resource Utilization Questionnaire | 3 months
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnoses and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those relating to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.
Healthcare Resource Utilization Questionnaire | 6 months
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnoses and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those relating to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.
Client Satisfaction Questionnaire (CSQ-8) | 1 week
  Intervention participants only. An 8-item scale that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction.
CBT Skills Questionnaire (CBTSQ) | 3 months
  Intervention participants only. A 16-item maternal-report measure designed to assess cognitive and behavioural skills acquisition. Each item is scored on a 5-point scale, and total scores range from 16-80. Higher cognitive restructuring and behavioural activation scores predict reduction of overall psychiatric symptoms and depression.
CBT Skills Questionnaire (CBTSQ) | 6 months
  Intervention participants only. A 16-item maternal-report measure designed to assess cognitive and behavioural skills acquisition. Each item is scored on a 5-point scale, and total scores range from 16-80. Higher cognitive restructuring and behavioural activation scores predict reduction of overall psychiatric symptoms and depression.
Working Alliance Inventory (WAI-SR) | 1 week
  Intervention participants only. A 12-item maternal-report measure that assesses three aspects of therapeutic alliance:(1) agreement on the tasks of therapy, (2) agreement on the goals of therapy and (3) development of an affective bond. Items are rated on a 5-point scale, and total scores range from 12-60 with higher scores indicating a better therapeutic alliance.
Mini International Neuropsychiatric Interview - Major Depressive Disorder Module | 3 months
  10-15 minute structured psychiatric interview will assess current psychiatric syndromes in participants by telephone at baseline to assess study eligibility. The MINI will be conducted again at 3 and 6 months to assess change in psychiatric symptoms over the study period.
Mini International Neuropsychiatric Interview - Major Depressive Disorder Module | 6 months
  10-15 minute structured psychiatric interview will assess current psychiatric syndromes in participants by telephone at baseline to assess study eligibility. The MINI will be conducted again at 3 and 6 months to assess change in psychiatric symptoms over the study period.
Estimate Treatment effect - Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  Estimate treatment effect of primary outcome for later RCT - The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score ≥13 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change.
Group cohesion - Therapeutic Factors Inventory - 8 item | 1 week
  Measured using the Therapeutic Factors Inventory-8 item that measures instillation of hope, secure emotional expression, awareness of relational impact and social learning. Items are scored on a likert-scale ranging from 1-7. Higher scores indicate a more cohesive group.
Development and testing of treatment fidelity measure | 12 weeks
  The fidelity with which the PHNs deliver the 1-Day CBT Workshop will be assessed using measures of adherence and competence. For this pilot study, adherence and competence measures will be developed and tested for use in a later RCT. Each workshop will be audio-recorded and trained raters will rate the adherence to the workshop model and competence with which the PHNs deliver the workshops.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Layton H, Campbell M, Huh K, Mansoor A, Serrano-Lomelin J, Brown JSL, Bieling PJ, Van Lieshout RJ. Public Health Nurse-Delivered 1-Day Cognitive Behavioral Therapy-Based Workshops for Treating Postpartum Depression: A Pilot Randomized Controlled Trial. J Clin Psychiatry. 2025 Apr 30;86(2):24m15712. doi: 10.4088/JCP.24m15712. PMID 40315102